CLINICAL TRIAL: NCT04596982
Title: Evaluation of Predictive Factors for Right Ventriculaire Dysfunction Post Implantation of Left Mono Ventricular Assistance in Patients in Cardiogenic Shock Under Veno Arterial ECMO
Brief Title: Evaluation of Predictive Factors for Right Ventriculaire Dysfunction
Acronym: ECPELLA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200528
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Right Ventriculaire Dysfunction
Keywords: ECMO, Right ventricule failure, Impella, circulatory support

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Placement of IMPELLA® — ultrasound and hemodynamic parameters of patients in order to establish a predictive score for right-sided dysfunction after placement of IMPELLA®

SUMMARY:
An observational study of patients in cardiogenic shock under veno-arterial ECMO is designed to describe the clinical, ultrasound and hemodynamic parameters of these patients and to establish a predictive score for right-sided dysfunction in a patient within 48 hours of ECMO withdrawal after placement of IMPELLA®.

DETAILED DESCRIPTION:
Therapeutic innovations in the field of heart failure are constant and have improved the prognosis and quality of life of patients. For those suffering from end-stage heart failure, heart transplantation remains the main therapeutic resource, but on the one hand the number of available grafts is insufficient compared to the number of transplant candidates, and on the other hand heart transplantation is accompanied by risks of rejection, infections and cancers, with a current median survival of 12 years .

For these reasons, in selected patients, a Left Ventricular Assist Device (LVAD) may be a bridge to transplantation or a way to improve the duration and quality of life of patients without a transplant project (destination therapy). Currently, about half of all heart transplants performed internationally are done in patients with left monoventricular assist, and in 2017 43% of implanted LVAD patients were in destination therapy.

For this reason, this observational study aims to describe the clinical, ultrasound and hemodynamic parameters of these patients and to establish a predictive score for right-sided dysfunction in a patient during the 30-day follow-up.

More precisely, during this study we will compare the clinical, ultrasound and hemodynamic parameters of these patients in order to establish a predictive score for right-sided dysfunction during :

* 48 hours on ECMO and IMPELLA (after IMPELLA® placement)
* 48 hours on IMPELLA alone following ECMO withdrawal.
* 48 hours under left monoventricular assistance
* At day 7 of the follow-up
* At day30 of the follow-up Patients who develop right heart failure within 48 hours of ECMO withdrawal after IMPELLA® placement will be compared to patients without right heart failure on demographic, clinical, history, treatment history, and cardiac echo and hemodynamic data at admission.

ELIGIBILITY:
Inclusion Criteria:

1. - Patient over 18 years of age
2. - Patient under ECMO hospitalized in the medical intensive care unit or the surgical intensive care unit of the Groupement hospitalier Pitié-Salpêtrière, not weaned from ECMO, in whom it was decided at the multidisciplinary collegial meeting on assistance-transplantation to set up an IMPELLA before the implantation of left monoventricular assistance.
3. - Patient who received informed information about the study and did not express opposition to participation in the research.

   Special Cases :

   o For patients who are unable to express their non-opposition, the investigator may request that of a relative of the patient.

   or For patients under guardianship, their non opposition must be obtained in the presence of the guardian.

   or For patients under guardianship, it is the legal guardian's non opposition that will be requested.

   The modalities of information and obtaining the non opposition will be reported in the patient's medical file.
4. - Patient affiliated or entitled to a French social security system -

Exclusion Criteria:

1. - SAPS-II Score > 90 (Simplified Acute Physiology Score (SAPS-II) at Inclusion
2. - Subject deprived of liberty by judicial decision
3. - Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients consecutively admitted to the cardiac medical and surgical intensive care units having : venoartrial ECMO and in whom the implantation of an assistance by IMPELLA is decided while waiting for the implantation of a left monoventricular assistance
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Absence of right heart failure or failure to withdraw ECMO due to right heart failure after placement of IMPELLA®. | Within 48 hours of ECMO withdrawal after placement of IMPELLA®
  The definition of right heart failure as defined by the INTERMACS takes into account the evolution of hemodynamic parameters during the 14 days following the implantation of the left monoventricular assist and is therefore not adapted to the situation of patients on veno-arterial ECMO who are going to have an IMPELLA for the purpose of ECMO weaning.

SECONDARY OUTCOMES:
Occurrence of severe right heart failure as defined by INTERMACS following implantation of left monoventricular assist | During all the follow-up 30 days
  Association of PVC > 16 mmHg and :
  * Continuation of inotropes or inhaled NO for more than 14 days. or
  * A right circulatory assistance at any time after the implantation of the LVAD or
  * Death related to right heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No